CLINICAL TRIAL: NCT04549662
Title: The HepatoPancreaticoBiliary Resection Arginine Immunomodulation (PRIMe) Trial: A Randomized Phase II Trial of the Impact of Perioperative Immunomodulation on Immune Function Following Resection for HepatoPancreaticoBiliary Malignancy
Brief Title: The HepatoPancreaticoBiliary Resection Arginine Immunomodulation (PRIMe) Trial
Acronym: PRIMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Enhanced Medical Nutrition (Industry); Sunnybrook Health Sciences Centre Clinical Research Grant Competition (Unknown); Sunnybrook Health Sciences Centre AFP Innovation Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 076-2017
Record Dates: First submitted 2020-08-14; First posted 2020-09-16 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-10

CONDITIONS: Hepatopancreaticobiliary (HPB) Malignancy; Surgery
Keywords: immunomodulation; omega-3 fatty acids; arginine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Powdered formula containing whey protein and arginine (Active A) and lipid bolus containing omega 3 fatty acids. Participants will mix the powder (Active A) with 250 mL of water and drink the formula 3 times per day for 5 days. Each drink will be followed by consuming 1 tsp of the lipid bolus. This will be done for 5 days prior to the operation and for 5 days after the operation.
  Interventions: Dietary Supplement: Active A; Dietary Supplement: Lipid bolus
- Group B (Active Comparator): Powdered formula containing whey protein and arginine (Active A) and placebo oil. Participants will mix the powder (Active A) with 250 mL of water and drink the formula 3 times per day for 5 days. Each drink will be followed by consuming 1 tsp of the lipid bolus. This will be done for 5 days prior to the operation and for 5 days after the operation.
  Interventions: Dietary Supplement: Active A; Dietary Supplement: Placebo oil
- Comparator (Placebo Comparator): Powdered formula containing whey protein (Active B) and placebo oil. Participants will mix the powder (Active B) with 250 mL of water and drink the formula 3 times per day for 5 days. Each drink will be followed by consuming 1 tsp of the lipid bolus. This will be done for 5 days prior to the operation and for 5 days after the operation.
  Interventions: Dietary Supplement: Active B; Dietary Supplement: Placebo oil

INTERVENTIONS:
Dietary Supplement: Active A — Powdered formula containing whey protein and arginine
  Arms: Group A; Group B
Dietary Supplement: Active B — Powdered formula containing whey protein
  Arms: Comparator
Dietary Supplement: Lipid bolus — Omega-3 fatty acids
  Arms: Group A
Dietary Supplement: Placebo oil — Control placebo oil that does not contain omega-3 fatty acids
  Arms: Comparator; Group B

SUMMARY:
This is a randomized controlled blinded superiority trial to evaluate the impact of perioperative immunosupplementation on immune function following resection for hepatopancreaticobiliary (HPB) malignancy.

DETAILED DESCRIPTION:
This is a 1:1:1 randomized controlled blinded superiority trial to evaluate the impact of perioperative immunosupplementation on immune function following resection for hepatopancreaticobiliary (HPB) malignancy. Two variations of immunosupplementation will be compared to control nutritional supplement containing whey protein with an additional teaspoon (tsp) of placebo oil. These variations will be 1) a powdered formula containing whey protein and arginine (Active A) with an additional tsp of lipid bolus containing omega-3 fatty acids, and 2) a powdered formula containing whey protein and arginine (Active A) with an additional tsp of placebo oil which does not contain omega-3 fatty acids. The control nutritional supplement will be a powdered formula containing whey protein with an additional tsp of placebo oil.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and over at time of diagnosis
* Resectable presumed liver, pancreas, or bile duct malignancy (i.e., liver metastases, HCC, cholangiocarcinoma, pancreatic or periampullary adenocarcinoma, NETs)as determined by surgeon in clinic
* Anticipated hospital stay at least three days post-surgery
* Ability to tolerate oral intake and comply with protocol requirements

Exclusion Criteria:

* Documented significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids, azathioprine, cyclosporin A). Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<7.5 mg daily)
* Subjects with resting hypotension (BP <90/50 at rest)
* History of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis
* Serious, active, intercurrent chronic or acute illness, or other active illness considered by the investigator as an unwarranted high risk for an investigational product
* Active infection of any site and/or active herpes requiring ongoing treatment
* Known pregnancy or nursing mothers
* Subjects with an allergy to the nutritional supplement or comparator including milk, fish and/or shellfish allergies
* Subjects with religious or other objections to consuming fish or shellfish
* Subjects with severe asthma defined as asthma not controlled with inhaled corticosteroids and additional controllers or by oral corticosteroid treatment (arginine can cause allergic response or make swelling in airways worse)
* Subjects with a known inherited guanidinoacetate methyltransferase deficiency (due to an inability to convert arginine to creatine)
* Subject with known current liver cirrhosis
* Subjects with documented myocardial infarction or life-threatening arrhythmia
* Subjects with known current cardiac failure or coronary artery disease causing unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Natural killer (NK) cell killing | Post-operative day 1 (Day 1) as compared to baseline (pre-operative)
  Reduction in NK cell killing as measured on post-operative day one (POD1) as compared to baseline (pre-operative) between the control and experimental cohorts. Nutritional supplementation will be considered effective at reducing postoperative NK cell dysfunction if there is a 50% or greater improvement in postoperative suppression of NK cell cytotoxicity (reduction of 27% from baseline).

SECONDARY OUTCOMES:
Secondary immune function outcomes: Immune cell subsets | Day of surgery to 30-days after surgery
  Flow cytometric analysis of different immune cell subsets to compare their proportions at all time points.
Secondary immune function outcomes: NK cell activating and inhibitory receptors | Day of surgery to 30-days after surgery
  Flow cytometric characterization of NK cell activating and inhibitory receptors to assess whether they are affected by immunosupplementation.
Secondary immune function outcomes: amino acid levels | Day of surgery to 30-days after surgery
  Systemic blood levels of amino acids will be measured via liquid chromatography-mass spectrometry protein card analysis.
Incidence of pancreatic fistula | Day of surgery to 90-days after surgery
  Pancreatic fistula of International Study Group on Pancreatic Fistula (ISGPF) Grade B & C (i.e. clinically significant) will be diagnosed clinically.
Postoperative wound complication and surgical site infection | Day of surgery to 90-days after surgery
  Wound complications including dehiscence and infection will be diagnosed clinically.
Length of stay | Day of surgery to day of discharge after surgery, assessed until day of discharge after surgery occurs
  Length of stay will be measured as number of days from admission to discharge.
90-day postoperative complications (Clavien-Dindo 3-5) | Day of surgery to 90-days after surgery
  Postoperative complications with Clavien-Dindo Grades 3-5 (i.e. requiring procedural intervention or ICU admission, or causing death) will be recorded.
90-day postoperative mortality | Day of surgery to 90-days after surgery
  The incidence of readmission within 90 days of surgery will be recorded as the number of days associated with each re-admission.
  Death within 90 days of surgery will be considered complications of the surgery.
Incidence of liver insufficiency | Day of surgery to 90-days after surgery
  Posthepatectomy liver failure of International Study Group of Liver Surgery (ISGLS) Grade B & C (i.e. clinically significant) will be diagnosed clinically

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Behman R, Auer RC, Bubis L, Xu G, Coburn NG, Martel G, Hallet J, Balaa F, Law C, Bertens KA, Abou Khalil J, Karanicolas PJ. Hepatopancreaticobiliary Resection Arginine Immunomodulation (PRIMe) trial: protocol for a randomised phase II trial of the impact of perioperative immunomodulation on immune function following resection for hepatopancreaticobiliary malignancy. BMJ Open. 2024 Apr 5;14(4):e072159. doi: 10.1136/bmjopen-2023-072159. PMID 38580363